CLINICAL TRIAL: NCT06594068
Title: PRIMULA Lac (Prospective Registry Investigating Maternal, Infant, and Lactation Outcomes in Anifrolumab Users): The AstraZeneca Lactation Study for Anifrolumab
Brief Title: Prospective Registry Investigating Maternal, Infant, and Lactation Outcomes in Anifrolumab Users
Acronym: PRIMULA Lac
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3461R00052
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Chronic autoimmune disease; Immunosuppressants; Corticosteroids; Human monoclonal antibody (IgG1ƙ mAb); Post Marketing Requirements (PMR) study
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anifrolumab (Experimental): Lactating individuals 18 years of age or older receiving anifrolumab therapeutically who provide consent to participate will be included in the study. Milk collection will occur at a series of 14 timepoints, 1 pre-dose (spot) and 13 post-dose: Day 1 [0-4 hours, 4-8 hours, 8-12 hours, 12-18 hours, 18-24 hours], Day 3 [48 hours, spot], Day 4 (spot), Day 6 (spot), Day 8 (spot), Day 12 (spot), Day 16 (spot), Day 22 (spot), and Day 29 (prior to next dose, spot). Maternal serum will be collected Day 1 (pre-dose and 0-4 hours post-dose), Day 12, and approximately Day 29 (immediately preceding subsequent dose). Infant serum will be collected on approximately Day 30 following the next dose and after 24 hours of breast feeding.
  Interventions: Drug: Anifrolumab

INTERVENTIONS:
Drug: Anifrolumab — Anifrolumab is a human monoclonal antibody that binds to subunit 1 of the type 1 interferon receptor, which was developed based on the evidence supporting the role of type 1 interferon pathway in SLE (Furie 2017). Clinical trial evidence from TULIP 1 and TULIP 2 have showed that monthly intravenous administration of anifrolumab led to a higher percentage of patients with a response, assessed with the British Isles Lupus Assessment Group-based Composite Lupus Assessment, compared with patients receiving placebo (Furie 2019; Morand 2020). Moreover, the phase II MUSE study showed that administration of anifrolumab resulted in substantially reduce disease activity, as measured by the SLE Responder Index, compared to patients receiving placebo (Furie 2017). These data resulted with applications to the FDA and the EMA, leading to approval by them in July 2021 and February 2022, respectively, for the treatment of adult patients with moderate to severe SLE who are receiving standard therapy.

SUMMARY:
Prospective Registry Investigating Maternal, Infant, and Lactation Outcomes in Anifrolumab Users (PRIMULA Lac) is a Post Marketing Requirements (PMR) study designed to fulfill the FDA post-marketing requirements. The study will collect data about the presence of anifrolumab in human breast milk and serum (maternal and infant) among lactating individuals who receive anifrolumab therapeutically.

DETAILED DESCRIPTION:
PRIMULA Lac is an open-label, open enrollment, post marketing study to assess concentrations of anifrolumab in breast milk and serum in lactating individuals who are receiving anifrolumab therapeutically, and to evaluate exposure on the breastfed infant. Milk collection will occur at a series of 14 timepoints. Maternal serum will be collected Day 1 (pre-dose and 0-4 hours post-dose), Day 12, and approximately Day 29 (immediately preceding subsequent dose). Infant serum will be collected on approximately Day 30 following the next dose and after 24 hours of breast feeding. Maternal and infant adverse events (AEs) will be actively collected for the duration of the study. Total duration of participation for each participant will be approximately 1 month. The objective of this lactation study is to assess presence of anifrolumab in breast milk and serum (maternal and infant) among lactating individuals who receive anifrolumab therapeutically and to evaluate exposure in the breastfed infant. This is a Post Marketing Requirements (PMR) study designed to fulfill the FDA post-marketing requirements.

ELIGIBILITY:
Inclusion Criteria:

Maternal:

1. 18 years or older
2. Signed informed consent to participate
3. Diagnosis of moderate/severe SLE
4. Ongoing treatment with anifrolumab
5. Has reached or will reach steady state (~85 days postpartum, at least 3 consecutive previous doses during the post-partum period) with anifrolumab by the time of study Day 1 (pre-dose milk collection)1
6. Established lactation in the index post-partum period (breastfeeding or pumping for at least 4 weeks at time of Day 1 visit to ensure mature milk production)
7. Willing to breastfeed or pump regularly during the study period to maintain milk supply and exclusively pump breast milk for the 24-hour period of breast milk collection on Day 1 post IV dose.
8. Plans to continue feeding infant breast milk at least throughout the duration of the study and is not weaning
9. Must be exclusively breast milk-feeding their infant (or if not exclusively breast milk-feeding, not providing more than 1 supplemental bottle of formula per day) at the time of enrollment and throughout the study period
10. Agrees to use only lanolin nipple cream during the sampling period

Infant:

1. Gestational age at delivery ≥32 weeks
2. Birthweight > 10th percentile
3. Weight > 10th percentile at the time of enrollment

Exclusion Criteria:

Maternal:

1. Received any investigational compound or approved biologic or biosimilar within 30 days or 5 half-lives (whichever is longer) prior to enrollment in the study
2. Diagnosis of lupus nephritis in the last 12 months5
3. History of breast implants, breast augmentation, or breast reduction surgery that significantly impacts breastfeeding or collection of milk from 1 or both breasts
4. History of malignancy in the last 10 years
5. History of mastectomy
6. Evidence of mastitis or any other significant active infection at Day 1 (pre-dose)

Infant:

1. Any abnormality noted or clinically significant medical condition, including cardiac, pulmonary, and liver disease, glucose instability, or active infection at the time of screening that, in the opinion of the investigator, may make implementation of the protocol or interpretation of the trial difficult or would put the infant participant at risk by participating in the study

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Area under the milk concentration-time curve during a dosing interval | Approximately 30 days
  Area under the milk concentration-time curve during a dosing interval is a component used to assess pharmacokinetic (PK) of anifrolumab in milk of lactating individuals. Milk PK parameters of anifrolumab will be derived using non-compartmental analysis methods and will be determined using the concentration-time data for all evaluable participants included in the PK population
Area under the milk concentration-time curve from time 0 to last quantifiable concentration | Approximately 30 days
  Area under the milk concentration-time curve from time 0 to last quantifiable concentration is a component used to assess PK of anifrolumab in milk of lactating individuals. Milk PK parameters of anifrolumab will be derived using non-compartmental analysis methods and will be determined using the concentration-time data for all evaluable participants included in the PK population
Average milk concentration at steady state | Approximately 30 days
  Average milk concentration at steady state is a component used to assess PK of anifrolumab in milk of lactating individuals. It will be calculated dividing "Area under the milk concentration-time curve during a dosing interval" by the dosing interval for anifrolumab
Observed milk concentration at end of dosing interval | Approximately 30 days
  Observed milk concentration at end of dosing interval is a component used to assess PK of anifrolumab in milk of lactating individuals. Milk PK parameters of anifrolumab will be derived using non-compartmental analysis methods and will be determined using data for all evaluable participants included in the PK population
Maximum observed milk concentration | Approximately 30 days
  Maximum observed milk concentration is a component used to assess PK of anifrolumab in milk of lactating individuals. Milk PK parameters of anifrolumab will be derived using non-compartmental analysis methods and will be determined using data for all evaluable participants included in the PK population
Time of maximum concentration | Approximately 30 days
  Time of maximum concentration is a component used to assess PK of anifrolumab in milk of lactating individuals. Milk PK parameters of anifrolumab will be derived using non-compartmental analysis methods and will be determined using data for all evaluable participants included in the PK population

SECONDARY OUTCOMES:
Total amount of drug excreted in milk over 24 hours | Day 1
  Variable used to assess total amount of drug excreted in milk of lactating individuals. Total amount of drug excreted in milk (mg) over 24 hours calculated as: Σ(total drug concentration in each milk collection x milk volume in each milk collection)
Fraction of dose excreted in milk | Day 1
  Variable used to assess fraction of anifrolumab dose excreted in milk of lactating individuals. Fraction of dose excreted in milk, calculated as (Total amount of drug excreted in milk over 24 hours)/Administered dose
Maternal serum pharmacokinetic (PK) concentrations | Maternal serum will be collected Day 1 (pre-dose and 0-4 hours post-dose), Day 12, and approximately Day 29 (immediately preceding subsequent dose)
  Variable used to assess maternal serum pharmacokinetic (PK) concentrations
Estimates of infant exposure | Infant serum will be collected on approximately Day 30 following the next dose and after 24 hours of breast feeding
  Variable used to assess infant anifrolumab exposure (daily infant dosage; relative infant dosage; infant serum anifrolumab concentration)
Maternal and Infant adverse events (AEs) | Total duration of participation for each participant will be approximately 1 month; data collection is planned for approximately 3 years
  Collection of maternal and/or infant AEs during study period. AEs will be summarized by system organ class, preferred term, severity, and causal relationship to anifrolumab

CONTACTS AND LOCATIONS:
Overall Officials: Darin Brimhall, MD, Principal Investigator — PPD, Las Vegas, US
Locations (1):
- Research Site, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from
  AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/